CLINICAL TRIAL: NCT03857893
Title: Thermal Treatment of Vulvo-vaginal Atrophy (VVA) Using Novel Low-energy Dynamic Quadripolar Radio-Frequency (DQRF)
Brief Title: New Non-Hormonal Treatment by Radiofrequency for Vulvo-Vaginal Atrophy
Acronym: ViViA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was delayed due to the Covid 19 pandemic. The study was stopped prematurely due to a lack of efficiency (reported by the patients)
Sponsor: Serge Rozenberg (Other)
Collaborators: NOVAVISION GROUP S.P.A (Unknown); Jules Bordet Institute (Other); Erasme University Hospital (Other); Centre Hospitalier Universitaire Brugmann (Other); Hôpitaux IRIS Sud (Unknown)
Responsible Party: Sponsor-Investigator, Serge Rozenberg, Head of Gynecology Department, Centre Hospitalier Universitaire Saint Pierre
Organization: Centre Hospitalier Universitaire Saint Pierre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B076201938646
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Vulvo-vaginal Atrophy; Genitourinary Syndrome of Menopause
Keywords: Vulvo-vaginal atrophy; Dynamic Quadripolar Radio-Frequency; Menopause; Genitourinary syndrome of menopause

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group : pH-Cream (Active Comparator): Control Group will be only treated with a fixed amount (1g) of pH-cream (Cetomacrogol cream) to self-administered with a vaginal applicator for 12 weeks (one dose every three days and if deem necessary, additional doses can be applied and notified in the calendar provided).
  Interventions: Drug: pH-Cream
- Dynamic Quadripolar Radio-Frequency treatment (Experimental): Experimental Group will be treated with Dynamic Quadripolar Radio-Frequency (DQRF) (with Eva™ Device) for 8 weeks (+ 4 weeks). The Dynamic Quadripolar Radio-frequency sessions will involve -5 sessions (one every 14-21 days), if necessary External treatment (vulvar - will be applied before internal treatment for more comfort) : 10 minutes (5 minutes left side, 5 minutes right side), and Internal treatment (VVA, Vaginal Laxity, Mild-Stress Urinary Incontinence (SUI)): 20 minutes.
  In parallel, patients can also apply pH-cream (Cetomacrogol cream) (one dose of 1g) if they judge necessary but they are not allowed to use it during the seven days before radiofrequency session. If they use pH-cream, they must notify it in the calendar provided.
  Interventions: Device: Dynamic Quadripolar Radio-Frequency treatment; Drug: pH-Cream

INTERVENTIONS:
Device: Dynamic Quadripolar Radio-Frequency treatment — Novel low-energy "Dynamic Quadripolar Radio-frequency" thermal treatment through Eva™ Device. Eva™ Device combines both advanced VDR™ technology (Vaginal Dynamic Radiofrequency) and RSS™ (Radiofrequency Safely System) technology.
  Arms: Dynamic Quadripolar Radio-Frequency treatment
Drug: pH-Cream — 1g of Cetomacrogol cream (pH-cream) to self-administered with a vaginal applicator for 12 weeks (one dose every three days)
  Other Names: Cetomacrogol cream

SUMMARY:
Vulvo-Vaginal Atrophy (VVA) or Genitourinary Syndrome of Menopause (GSM) is a common and under-reported condition associated with decreased estrogenization of the vaginal tissue The aim of this study is to evaluate safety and efficacy of " Dynamic Quadripolar Radio-frequency" thermal treatment with Vaginal Dynamic Radio-frequency (VDR™) and Radio-frequency Safety System (RSS™) for the treatment of VVA and GSM in postmenopausal women who either present contra-indication for menopause hormone therapy, or are not willing to use Menopause Hormone Therapy (MHT) or have failed to be helped using MHT.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women suffering of Vulvo-Vaginal atrophy (VVA), included Breast Cancer survivors defined as having self-identified at least one mild to severe of the following symptoms:

  1. Vaginal dryness (none, mild, moderate or severe),
  2. Vaginal and/or vulvar irritation/itching (none, mild, moderate or severe),
  3. Vaginal pain associated with sexual activity (none, mild, moderate or severe)
* Postmenopausal women with VVA confirmed by at least one of the following criteria:

  1. A proportion of superficial cells ≤ 5% in the vaginal smear using a "Maturation Index"
  2. A vaginal pH > 5
* Postmenopausal women between 40 and 75 years of age (non hysterectomized or hysterectomized). Menopause will be assessed either by amenorrhea of > 1 year and / or by Follicle Stimulating Hormone (FSH) > 30 UI/L and estradiol (E2) < 20 pg/ml
* They must have either a contraindication to hormonal therapies, a failure of previous use of hormonal therapies (either systemic and/or local) or must have refused to take hormonal therapy.
* Willing to participate in the study and sign an informed consent.

Exclusion Criteria:

* Undiagnosed abnormal genital bleeding.
* The administration of any investigational drug within 30 days of screening visit.
* Endometrial hyperplasia at biopsy performed at screening or endometrial cancer.
* Use of estrogens/progestins products (vaginal, oral, pellet, transdermal....) in the 4 weeks to months (depending on the product used) prior study entry.
* Presence of severe medical disease or neurological disease or important co-morbidities.
* Other gynaecological malignancies.
* Recent vaginal surgery .
* A clinically relevant prolapse (Pelvic Organ Prolapse-Quantification System (POP-Q) ≤ 2)
* Current urinary tract or vaginal infection or recent sexually transmitted disease
* Anticoagulant treatment
* People with pacemakers and/or other implanted electrodes (Intra-Uterine Device (IUD) and surgical pelvic implants for sterilization are not considered as contraindication)
* Disabled people unable to communicate

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 53 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 12 (+4 weeks) of self-assessment of the most bothersome symptom dyspareunia, evaluated by a questionnaire | Up to 12 (+4 weeks) week after beginning of treatment
  The severity of dyspareunia recorded as none, mild, moderate or severe (score values of 0, 1, 2 or 3, respectively). Data obtained at baseline and week 12 (+4 weeks).
Change from baseline to week 12 (+4 weeks) of vaginal cell maturation (Maturation Index). | Up to 12 (+4 weeks) week after beginning of treatment
  The percentage of parabasal, superficial, intermediate cells will be determined from the vaginal smears collected during the study at baseline and week 12 (+4 weeks). The maturation index is the proportion of these 3 types of cells in each 100 cells counted on a smear.
Change from baseline to week 12 (+4 weeks) of vaginal pH | Up to 12 (+4 weeks) week after beginning of treatment
  A pH strip will be applied directly to the lateral wall of the vagina using forceps. The change in color of the pH indicator strip will be compared to the color chart for pH evaluation.Data obtained at baseline and week 12 (+4 weeks)

SECONDARY OUTCOMES:
Change from baseline to week 12 (+4 weeks) of the "Vaginal Health Index" (VHI) | Up to 12 (+4 weeks) week after beginning of treatment
  Evaluation of each of the four following signs of atrophy, which constitute together the Vaginal Health Index" (VHI). Vaginal Secretions, Vaginal Epithelial Integrity, Vaginal Epithelial Surface Thickness, Vaginal Color will be evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy and will be analyzed using the score values of 1, 2, 3 and 4, respectively. The visual evaluation of the vagina (petechiae, pallor, friability and dryness or redness in vaginal mucosa) will be assessed using the pictures by the physician blinded to the treatment. Data will be obtained at baseline and week 12 (+4 weeks).
Change from baseline to week 12 (+4 weeks) of the vulvovaginal symptoms | Up to 12 (+4 weeks) week after beginning of treatment
  The vulvovaginal symptoms will be evaluated by a 'vulvovaginal symptoms questionnaire" in postmenopausal women at baseline and week 12 (+4 weeks).
Change from baseline to week 12 (+4 weeks) in the two groups of the "Female Sexual Function Index (FSFI) | Up to 12 (+4 weeks) week after beginning of treatment
  The Female Sexual Function Index is measured by a questionnaire evaluating self-reported sexual functioning during the previous month. This includes 19 items grouped within six central domains: desire (items 1 and 2), arousal (items 3 to 6), lubrication (items 7 to 10), orgasm (items 11 to 13), global sexual and relationship satisfaction (items 14 to 16), and pain (items 17 to 19). Each domain was scored on a scale of 0 to 6 with lower scores indicating lower sexual functioning. A domain score of 0 indicated that the women reported no sexual activity. The individual domain scores were then totaled and multiplied by a predetermined factor to weight each domain equally.

CONTACTS AND LOCATIONS:
Overall Officials: Serge Rozenberg, MD,PhD, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (5):
- Belgium (5):
  - CHU Brugmann, Brussels
  - CHU Saint-Pierre, Brussels
  - Hôpital Erasme, Brussels
  - Hôpitaux Iris Sud, Brussels
  - Jules Institute Bordet, Brussels

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared and will be available on a website at the end of the study. The website where the data will be hosted, has not been yet decided.

REFERENCES:
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Erekson EA, Yip SO, Wedderburn TS, Martin DK, Li FY, Choi JN, Kenton KS, Fried TR. The Vulvovaginal Symptoms Questionnaire: a questionnaire for measuring vulvovaginal symptoms in postmenopausal women. Menopause. 2013 Sep;20(9):973-9. doi: 10.1097/GME.0b013e318282600b. PMID 23481118
- [Background] Bouchard C, Labrie F, Derogatis L, Girard G, Ayotte N, Gallagher J, Cusan L, Archer DF, Portman D, Lavoie L, Beauregard A, Cote I, Martel C, Vaillancourt M, Balser J, Moyneur E; VVA Prasterone Group. Effect of intravaginal dehydroepiandrosterone (DHEA) on the female sexual function in postmenopausal women: ERC-230 open-label study. Horm Mol Biol Clin Investig. 2016 Mar;25(3):181-90. doi: 10.1515/hmbci-2015-0044. PMID 26725467
- [Background] Vicariotto F, DE Seta F, Faoro V, Raichi M. Dynamic quadripolar radiofrequency treatment of vaginal laxity/menopausal vulvo-vaginal atrophy: 12-month efficacy and safety. Minerva Ginecol. 2017 Aug;69(4):342-349. doi: 10.23736/S0026-4784.17.04072-2. PMID 28608667
- [Background] Rozenberg S, Vandromme J, Antoine C. Postmenopausal hormone therapy: risks and benefits. Nat Rev Endocrinol. 2013 Apr;9(4):216-27. doi: 10.1038/nrendo.2013.17. Epub 2013 Feb 19. PMID 23419265
- [Background] Nappi RE, Kokot-Kierepa M. Women's voices in the menopause: results from an international survey on vaginal atrophy. Maturitas. 2010 Nov;67(3):233-8. doi: 10.1016/j.maturitas.2010.08.001. Epub 2010 Sep 9. PMID 20828948
- [Background] Melisko ME, Goldman ME, Hwang J, De Luca A, Fang S, Esserman LJ, Chien AJ, Park JW, Rugo HS. Vaginal Testosterone Cream vs Estradiol Vaginal Ring for Vaginal Dryness or Decreased Libido in Women Receiving Aromatase Inhibitors for Early-Stage Breast Cancer: A Randomized Clinical Trial. JAMA Oncol. 2017 Mar 1;3(3):313-319. doi: 10.1001/jamaoncol.2016.3904. PMID 27832260
- [Background] Kingsberg SA, Wysocki S, Magnus L, Krychman ML. Vulvar and vaginal atrophy in postmenopausal women: findings from the REVIVE (REal Women's VIews of Treatment Options for Menopausal Vaginal ChangEs) survey. J Sex Med. 2013 Jul;10(7):1790-9. doi: 10.1111/jsm.12190. Epub 2013 May 16. PMID 23679050
- [Background] Kendall A, Dowsett M, Folkerd E, Smith I. Caution: Vaginal estradiol appears to be contraindicated in postmenopausal women on adjuvant aromatase inhibitors. Ann Oncol. 2006 Apr;17(4):584-7. doi: 10.1093/annonc/mdj127. Epub 2006 Jan 27. PMID 16443612
- [Background] Hutchinson-Colas J, Segal S. Genitourinary syndrome of menopause and the use of laser therapy. Maturitas. 2015 Dec;82(4):342-5. doi: 10.1016/j.maturitas.2015.08.001. Epub 2015 Aug 12. PMID 26323234
- [Background] Baumgart J, Nilsson K, Evers AS, Kallak TK, Poromaa IS. Sexual dysfunction in women on adjuvant endocrine therapy after breast cancer. Menopause. 2013 Feb;20(2):162-8. doi: 10.1097/gme.0b013e31826560da. PMID 22990756
- [Background] Antoine C, Vandromme J, Fastrez M, Carly B, Liebens F, Rozenberg S. A survey among breast cancer survivors: treatment of the climacteric after breast cancer. Climacteric. 2008 Aug;11(4):322-8. doi: 10.1080/13697130802244422. PMID 18645698
- [Background] Antoine C, Liebens F, Carly B, Pastijn A, Rozenberg S. Safety of alternative treatments for menopausal symptoms after breast cancer: a qualitative systematic review. Climacteric. 2007 Feb;10(1):23-6. doi: 10.1080/13697130601176734. PMID 17364601
- [Background] Ameye L, Antoine C, Paesmans M, de Azambuja E, Rozenberg S. Menopausal hormone therapy use in 17 European countries during the last decade. Maturitas. 2014 Nov;79(3):287-91. doi: 10.1016/j.maturitas.2014.07.002. Epub 2014 Aug 4. PMID 25156453
- [Background] Goldstein SR, Bachmann GA, Koninckx PR, Lin VH, Portman DJ, Ylikorkala O; Ospemifene Study Group. Ospemifene 12-month safety and efficacy in postmenopausal women with vulvar and vaginal atrophy. Climacteric. 2014 Apr;17(2):173-82. doi: 10.3109/13697137.2013.834493. Epub 2013 Nov 23. PMID 23984673
- [Background] Rozenberg S, Pornel B, Koninckx PR, Palacios S, Christiansen C. Endometrium protection and acceptability of nasally administered continuously combined hormone therapy: a multicentre, multinational, double-blind trial in post-menopausal women evaluating three regimens of 17beta-estradiol and norethisterone when compared with an orally administered 17beta-estradiol norethisterone regimen. Hum Reprod. 2009 Jul;24(7):1739-47. doi: 10.1093/humrep/dep067. Epub 2009 Apr 7. PMID 19351658
- [Derived] Joris A, Di Pietrantonio V, Praet J, Renard K, Verduyn AC, Buxant F, Rozenberg S. Randomized trial: treatment of genitourinary syndrome of menopause using radiofrequency. Climacteric. 2024 Apr;27(2):210-214. doi: 10.1080/13697137.2024.2302425. Epub 2024 Jan 22. PMID 38251861